CLINICAL TRIAL: NCT01564498
Title: A Pilot Study of the Effects of Replacing Orange Carrots and White Potatoes With Purple Varieties, on Risk Factors for Cardiovascular Disease
Brief Title: Effects of Purple Vegetables on Cardiovascular Disease (CVD) Risk Factors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government)
Responsible Party: Principal Investigator, Kelly Anne Meckling, PhD, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012MeckPurpleVeg
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension; Hypercholesterolemia; Type II Diabetes; Obesity; Inflammation
Keywords: anthocyanins; antioxidant; polyphenols; bioavailability; cholesterol; insulin sensitivity; glucose tolerance; atherosclerosis; metabolic syndrome
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Diabetes Mellitus, Type 2; Obesity; Inflammation; Insulin Resistance; Atherosclerosis; Metabolic Syndrome | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- White potato (Placebo Comparator): Participants will consume 300-500 g of cooked white potatoes per day
  Interventions: Other: vegetable
- Purple Potato (Experimental): Participants will consume 300-500 g of cooked purple potato per day
  Interventions: Other: vegetable
- Orange carrots (Placebo Comparator): Participants will consume 200-300 g typical varieties of orange carrots during the intervention
  Interventions: Other: vegetable
- Purple Carrots (Experimental): Participants will consume 200-300 g raw purple carrots instead of orange carrots in the control arm
  Interventions: Other: vegetable

INTERVENTIONS:
Other: vegetable — 200-300 g raw carrots or 300-500 g cooked potatoes

SUMMARY:
The hypothesis is that richly coloured purple vegetables, rich in polyphenolic compounds including anthocyanins will have higher antioxidant and other biological activities, than more lightly coloured versions of these foods. Diets of human subjects will be modified to allow consumption of 200-300 g of raw carrots or cooked potatoes. Participants will be randomized to consume either orange or purple carrots, or white or purple potatoes. They will consume these diets for 12 weeks and bioavailability of polyphenolics will be examined as well as anthropometry and blood biochemistry for changes in risk factors associated with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* adult men and women 18-65 years of age
* must have a least one of the following risk factors associated with increased risk of type II diabetes and/or cardiovascular disease:

  * borderline high or hypertension or undergoing treatment for such
  * abnormal fasting blood glucose or undergoing treatment for such
  * overweight or obese
  * borderline high or high LDL-cholesterol or undergoing treatment for such
  * borderline low or low HDL-cholesterol
  * borderline high or high triglycerides or undergoing treatment for such

Exclusion Criteria:

* smokers, pregnant or nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Blood cholesterol | 12 weeks
  blood will be collected at baseline before the experimental foods are introduced and again 6 weeks into the intervention period and during the last week of the intervention (week 12)

SECONDARY OUTCOMES:
blood pressure | 12 weeks
  Participants will have their body weight and blood pressure taken at weekly counselling sessions
body composition | 12 weeks
  body composition will be measured in well hydrated subjects using bioelectric impedence analysis
insulin resistance | 12 weeks
  insulin resistance will be measured by way of an oral glucose tolerance test and collection of venous blood samples for the subsequent 3 hours on two occasions, baseline and during the last week of the intervention diet.
blood and urinary polyphenol metabolites | 12 weeks
  venous blood and urine will be collected to determine the metabolic profiles of polyphenolics in individual participants.
  Based on intake data, the bioavailability of the polyphenols in the foods will be estimated.
circulating biomarkers of cardiovascular disease and type II diabetes risk | 12 weeks
  Blood will be collected for measurement of multiple cytokines, growth factors and other blood biomarkers associated with these diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No